CLINICAL TRIAL: NCT06702410
Title: WHO Mental Health Gap Action Program (mhGAP) Delivered by Primary Care Workers for Improving Quality of Child Mental and Behavioral Disorders Services: A Hybrid Effectiveness-implementation Cluster Randomized Controlled Trial
Brief Title: WHO Mental Health Gap Action Program (mhGAP) for Improving Child Mental and Behavioral Disorder Service Quality in China
Acronym: mhGAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wen Chen, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-089; 20-389 (Other Grant/Funding Number: China Medical Board); 2022B1515020094 (Other Grant/Funding Number: Guangdong Outstanding Youth Fund)
Record Dates: First submitted 2024-11-20; First posted 2024-11-25 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Neurodevelopmental Disorders
Keywords: neurodevelopmental disorders; task shifting; evidence-based practice; implementation science; stepped wedge trial
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: This study use a stepped wedge design. Participants in the same kindergarten are defined as a cluster. The study includes four sequence, each sequence includes five clusters. Each Sequeces will transform into mhGAP-IG intervention as predominated order. Thus the study includes 20 clusters totally.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the adapted mhGAP-IG (Experimental): mhGAP-IG-based CMBDs mental health services (including screening, management and follow-up) delivered by trained kindergarten teachers
  Interventions: Behavioral: mental health gap action program intervention guide (mhGAP-IG)

INTERVENTIONS:
Behavioral: mental health gap action program intervention guide (mhGAP-IG) — The mhGAP-IG is an evidence-based intervention developed by WHO. It was designed for non-specialists to scale up high quality mental health services. Although more than 90 countries worldwide have implemented mhGAP-IG, this study is the first to evaluated if it works for scaling up CMBDs services in China. Investigators have cultrually adapted the mhGAP-IG according Chinese context.

SUMMARY:
The goal of this clinical trial is to learn if the adapted mhGAP intervention guide (mhGAP-IG) can improve quality of child mental and behavioral disorders (CMBDs) services in China. It will also learn about the implementation of the mhGAP-IG delivered by kindergarten teachers. The main questions it aims to answer are:

* Does the adapted mhGAP-IG reduce the symptom severity among children with CMBDs between two and sis years old?
* Does the adapted mhGAP-IG reduce psychological distress among caregivers of children with CMBDs?
* Does the adapted mhGAP-IG improve mental and behavioral health serivces capacity among kindergarten teachers in China?
* How is the feasibility, acceptablity, and what are barriers and facilitators of implementation?

Researchers will compare the adapted mhGAP-IG to child healthcare as usual to see if the adapted mhGAP-IG can improve quality of child mental and behavioral disorders services in China.

Participants (kindergarten teachers) will:

* Complete questionnaires and scales at baseline and at 3-, 6-, 9- and 12- months of intervention;
* Receive mhGAP-based trainings;
* Deliver long-term child mental and behavioral disorders services (including screenings, referals, follow-up, and physcosocial interventions) to children with CMBDs.

Participants (children/caregivers) will:

* Complete questionnaires and scales at baseline and at 3-, 6- and 12- months of intervention.
* Accept long-term CMBDs management (including screenings, referals, follow-up management, and physcosocial interventions) from mhGAP-trained kindergarten teachers.

DETAILED DESCRIPTION:
Background: Globally, child mental and behavioral disorders (CMBDs) have a high disease burden. The quality of CMBDs services in China, and in many low- and middle-income countries (LMICs), is limited due to the shortage of mental health providers trained to deliver evidence-based clinical care for this population. The WHO Mental Health Gap Action Program Intervention Guide (mhGAP-IG)is an evidence-based training for non-specialist mental health providers in LMICs.

Overall goal: Using a hybrid Type I trial design, To evaluate the effectiveness and implementation of the adapted mhGAP-IG at kindergartens in Guangdong province, China.

Methods: The effectiveness and implementation of the adapted mhGAP-IG will be tested in a stepped-wedge cluster randomized controlled trial. The trail will recruit 20 kindergartens and 375 children in Zhongshan City. Kindergartens will be randomly and subsequently enrolled at regular intervals (steps). At each step, kindergarten teachers will receive the mhGAP-IG training and then cross over from the control condition (providing child mental and behavioral disorders services as usual) to the intervention condition (providing child mental and behavioral disorders services under the adapted mhGAP-IG).

Outcome measures:Symptom severity of CMBDs measured by the Strengths and Difficulties Questionnaire is set as the primary outcome. Implementation measurements will cover the five domains of the Reach, Effectiveness, Adoption, Implementation, Maintenance (RE-AIM) framework.

Implications: This project will provide additional evidence of the effectiveness of the mhGAP-IG in improving quality of CMBDs services. The lessons learned from this project can aid in scaling the training to other regions of China and LMICs.

ELIGIBILITY:
1. Eligibility criteria for children/caregivers

   Inclusion Criteria:
   * Aged 2-6 years;
   * Screened positive by the mhGAP-IG screening tool;
   * Will stay in Zhongshan City for the next one year.

   Exclusion Criteria:
   * Co-morbid physical or mental conditions requiring inpatient hospitalization;
   * Currently or in the past six months received CMBDs services provided by specialized mental health workers;
   * Deafness or blindness in the child or caregivers;
   * Not available or unwilling to participate in the trial.
2. Eligibility criteria for kindergarten teachers

Inclusion Criteria:

* Have one or more years of work experience in the selected kindergartens
* Be available to participate in the mhGAP training.

Exclusion Criteria:

* Have received the mhGAP training before;
* Have arrangements requiring long-term leave from work in the next one year;
* Unwilling to participate in the trial.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 375 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Symptom severity of CMBDs assessed by Strengths and Difficulties Questionnaire (SDQ) | baseline and 3-, 6- and 12- months of intervention
  A total score ranges from 0 (lowest distress) to 60 (highest distress) and higher scores of SDQ indicate the worse symptom.
Developmental domain scores measured by Ages and Stages Questionnaire (ASQ) | baseline and 3-, 6- and 12- months of intervention
  Developmental domain scores derived from ASQ. The ASQ consists of a series of questionnaires specifically designed for children at different months of age. The total score range varies depending on the questionnaire for each age group, but higher scores consistently indicate better development within a particular domain.

SECONDARY OUTCOMES:
Caregivers' psychological distress assessed by the Parenting Stress Index-Short Form (PSI-SF) | baseline and 3-, 6- and 12- months of intervention
  A total score ranges from 7 (lowest distress) to 28 (highest distress).
Mental health action competence among kindergarten teachers measured by the Chinese version of Mental Health Action Competence (MHAC) Scale. | baseline and 3-, 6-, 9-, and 12- months of intervention
  A total score ranges from 4 (lowest self-reported competence) to 64 (highest lowest self-reported competence).
Kownledge level on providing CMBDs services among kindergarten teachers measured by the knowledge questionnaire form the mhGAP-IG | baseline and 3-, 6-, 9-, and 12- months of intervention
  The questionnaire consists of a series of multiple-choice questions regarding the assessment, management, and follow-up of CMBD. Each correct answer is awarded one point, while incorrect answers receive no points. A higher total score indicates a greater level of knowledge.
Efficacy score among kindergarten teachers measured by the Chinese short form Teacher Efficacy Scale (TSE). | baseline and 3-, 6-, 9- and 12- months of intervention
  The TSE consists of measures for efficacy for instructional strategies, for classroom management, and for student engagement. Both total score or subscale score can derived from TSE, and higher score indicates a greater level of efficacy.

OTHER OUTCOMES:
Adoption and maintainance of the intervention measured by the proportion of targeted teahcers who attended the mhGAP trainings, the screenings rate in each class/kindergarten, the referal rate and follow-up rate in each kindergarten. | baseline, 3-, 6-, 9-, 12-months of intervention.
  One teacher in each class will be recruited, so that the number of targeted teacher equals to the number of classes in a kindergarten. The screening rate in class will be calculated as the number of children screened in a class divided by the total number of children in the class. The screening rate in class will be calculated as the number of children screened in a kindergarten divided by the total number of children in the kindergarten. The referal rate equals to the number of children be refered divided by the number of children screened positive. The follow-up rate equals to the number of children be followed divided by the number of children screened positive.
Number of children who are referred to hospital and diagnosed with CMBDs | From enrollment to 12 months of intervention
  The diagnosis will be made by clinical professionals in CMBDs

CONTACTS AND LOCATIONS:
Overall Officials: Wen Chen, PhD, Principal Investigator — Medical statistics, School of public health, Sun Yat-sen University
Locations (9):
- China (9):
  - Zhongshan Zhengfa Kindergarten, Zhongshan, Guangdong
  - Zhongshan Xiaolan Huasheng Kindergarten, Zhongshan, Guangdong
  - Zhongshan Dongfeng Deshan Kindergarten, Zhongshan, Guangdong
  - Zhongshan Huangpu Boya Oriental Pearl Kindergarten, Zhongshan, Guangdong
  - First Kindergarten in Zhongshan Torch High-Tech Industrial Development Zone, Zhongshan, Guangdong
  - Third Kindergarten in Zhongshan Torch High-Tech Industrial Development Zone, Zhongshan, Guangdong
  - Xiao Yin Kindergarten in Zhongshan Torch High-Tech Industrial Development Zone, Zhongshan, Guangdong
  - Zhangjiabian Kindergarten in Zhongshan Torch High-Tech Industrial Development Zone, Zhongshan, Guangdong
  - Shaxi Xin Shimen Kindergarten in Zhongshan City., Zhongshan, Guangdong

IPD SHARING:
Plan to Share IPD: No